CLINICAL TRIAL: NCT05866874
Title: Continuous Monitoring of Vital Signs for Improved Phenotyping of Perioperative Myocardial Infarction/Injury After Noncardiac Surgery in High Risk Patients: PMI-VITAL
Brief Title: Monitoring of Vital Signs for Phenotyping of Perioperative Myocardial Infarction/Injury After Noncardiac Surgery
Acronym: PMI-VITAL
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: PMI VITAL; 2021-02274 (Other: BASEC)
Record Dates: First submitted 2023-05-10; First posted 2023-05-19 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Perioperative Myocardial Infarction; Perioperative Myocardial Injury
Keywords: Perioperative myocardial injury/infraction; Myocardial ischemia/diagnosis; Myocardial ischemia/epidemiology; Perioperative complications/diagnosis; PMI
MeSH Terms: conditions — Myocardial Ischemia; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational prospective cohort study is to learn about the pathophysiology of perioperative myocardial infarction/injury in high-risk patients undergoing major non-cardiac surgery.

Participants will:

* Wear wearable device (Basler Band) for up to seven days after the operation or until hospital discharge
* Provide three blood samples. A venous specimen of blood (25 mL) will be collected preoperatively and on postoperative days 1 and 2.
* Be contacted to answer a questionnaire one year after the surgery.

DETAILED DESCRIPTION:
Background:

With over 300 million surgical procedures performed annually, surgery and anaesthesia provide major medical value to patients, especially in resource-rich countries like Switzerland with about 900.000 procedures done per year. Demand for surgery is expected to further increase in the coming years due to the aging of the population and the availability of novel less invasive surgical procedures making even elderly patients with extensive comorbidities possibly eligible for surgery.

Perioperative myocardial infarction/injury (PMI) has been identified as a major contributor to perioperative mortality. First studies estimated that PMI is a major contributor to 34-42% of all deaths following noncardiac surgery within 30 days. Recent research by several groups including ours has highlighted that PMI is not a homogenous disease entity, but seems to comprise several underlying pathophysiologies. These include type I myocardial infarction due to atherothrombosis, type II myocardial infarction due to myocardial oxygen supply-demand mismatch, tachyarrhythmias, acute heart failure, and PMI due to primarily extra-cardiac disorders such as severe sepsis, stroke, or pulmonary embolism. Unfortunately, the underlying pathophysiology of PMI remains unknown in many patients. This is among other things due to incomplete recording and documentation of patient vital signs including heart rate, blood pressure, and oxygen saturation e.g. in the postoperative period once patients leave the operating room. Identifying the underlying trigger of PMI is a prerequisite for causal therapy and prevention.

Objectives:

1. To continuously document and quantify the frequency and duration of tachyarrhythmia, bradycardia, hypotension, hypertension, and/or hypoxemia, that are not recorded and documented using the current clinical monitoring standards, but detected using continuous monitoring of vital signs using the wearable device (Basler Band) throughout the whole perioperative period.
2. To validate the diagnosis of PMI within a screening program in high-risk patients undergoing major noncardiac surgery with other troponin assays.
3. To evaluate the diagnostic and predictive utility of novel biochemical markers.
4. To technically validate intraoperative haemodynamic measurements of wearable device by comparing them to routinely obtained intraoperative haemodynamics.

Number of Participants:

We expect PMI to occur in 15-20% of patients. We expect 35% of cases to fall in the adjudication category of "cardiac, unknown" in first adjudication. Continuous vital signs and biomarkers are expected to allow to adjudicate ~33% of PMI from the category "unknown" to any of the other definite categories. Using a Chi-square test for final analysis, we calculate a needed sample size of approximately 125 PMI. With worst-case PMI-incidence of 15%, and a buffer of 5% additional cases to compensate for technical difficulties which are expected to arise with continuous monitoring, we require a total sample size of 875 patients included into the cohort.

Methodology:

After obtaining written informed consent, a venous specimen of blood (25 mL) is collected preoperatively and the patient will receive the wearable device. Further venous blood samples are withdrawn on postoperative days 1 and 2 (each 25 mL). As all patients will be included into the routine troponin screening implemented at the University Hospital Basel, blood draws will be coordinated with routine blood draws as far as possible. The wearable device will be worn until seven days after surgery or until hospital discharge.

Project duration for each patient will be approximately one week plus the answering of a questionnaire one year after the surgery.

Biobank:

One preoperative and two postoperative venous blood samples are collected into plastic tubes containing sodium citrate 1:10 (4.3 mL), heparin (4.7 mL), ethylenediaminetetraacetic acid (EDTA, 7.5 mL) and a clotting activator for serum diagnostics (7.5 mL). The biological material collected will be coded and stored on study site (or in the biobank of the University Hospital Basel) for an indefinite period of time. During this timeframe the collected biological material can be used for future, not yet further defined research projects.

Wearable device: Basler Band (MMT 278-1 Bracelet) The multi-sensor wearable devices (Basler Band) will be provided by Manufacture Modules Technologies (MMT). The Basler Band relies on the MMT-CW287 multisensor technology to simultaneously and unobtrusively detect up to 9 core body parameters, and convey the information to physicians in a secure and GDPR- compliant fashion. It includes sensors and algorithms to measure heart rate, heart rate variability, heart rhythm, respiration rate and activity.

For validating the quality of the Basler Band, additional devices were used to collect photoplethysmographic data and tested on a limited number of patients. All devices have CE-markings to ensure the compliance with safety standards for medical devices. Basler Band version 2 consists of a sensor from the PulseWatch Model D, manufactured and developed by the CSEM (Neuchâtel, Switzerland). Basler Band version 3 consists of a sensor from the epyGuard model which is manufactured and developed by epyMetrics AG.

ELIGIBILITY:
Inclusion Criteria:

* Patient eligible for routine PMI-screening
* Patient requiring hospitalisation with ≥ 2 overnight stays after surgery
* Age ≥ 40 years to ≤ 85 AND history of coronary artery disease (CAD), peripheral artery disease (PAD), cerebrovascular disease/stroke, insulin-dependent diabetes mellitus (IDDM), or chronic heart failure (CHF)
* Elective surgery
* Patients undergoing orthopaedic, traumatology, vascular, spinal, thoracic, neurosurgical, urological or visceral surgery
* Patient consent available

Exclusion Criteria:

* Patient's refusal
* Heart surgery, cardiac arrest, acute mycardial infarction (AMI), cardiac valve intervention, or cardiac catheter ablation within 14 days prior to surgery OR involvement of heart surgery at index surgery OR surgery planned on cardiopulmonary bypass
* Patients undergoing plastic/reconstructive, ophthalmologic, dental, hand surgery, or ear-nose-and-throat surgery
* Chronic renal failure on dialysis, unless undergoing renal transplant surgery
* Moderate to severe dementia
* Inclusion into study within the last year

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients that underwent a systematic approach to PMI detection at the hospital as clinical routine will be included.
Sampling Method: Probability Sample
Enrollment: 875 (Estimated)
Dates: Start 2022-09-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Perioperative myocardial infarction/injury (PMI) | 3 days after surgery
  PMI is defined as an absolute increase in high-sensitivity cardiac troponin (hs-cTn) of the 99th percentile of healthy individuals for the respective assay above baseline cTn-value or between two postoperative values if the preoperative value was missing.
  PMI will be further classified as type I myocardial infarction, type II myocardial infarction, or myocardial injury due to non-cardiac causes. Two independent cardiologists or anaesthesiologists will adjudicate all PMI cases.
Major adverse cardiac and cerebral events (MACCE) | 1 year
  MACCE is defined as a composite of all-cause death, acute myocardial infarction, acute heart failure (requiring admission to a hospital or intra-hospital transfer to the internal medicine or intensive care unit), clinically relevant arrhythmias (cardiac arrest, sustained ventricular tachycardia, atrioventricular (AV)-block III, high rate atrial fibrillation/flutter requiring treatment, bradycardia requiring pacemaker, or rhythmogenic syncope) and stroke/transient ischaemic attack within one year.
Postoperative atrial fibrillation (POAF) | During surgery and up to 7 days after surgery or until hospital discharge.
  POAF is defined as new-onset atrial fibrillation (AF) in the immediate postoperative period of duration/burden at least 30 minutes detected using continuous monitoring of vital signs using the wearable device (Basler Band), but not recorded and documented using the current clinical monitoring standards.
Documentation and quantification of the frequency and duration of tachyarrhythmia, bradycardia, hypotension, hypertension, and/or hypoxaemia. | During surgery and up to 7 days after surgery or until discharge.
  Frequency and duration of tachyarrhythmia, bradycardia, hypotension, hypertension, and/or hypoxaemia detected using continuous monitoring of vital signs using the "Basler Band" throughout the whole perioperative period, and use this information to characterise PMI.
  Major abnormalities will be defined as: hypotension (systolic blood pressure <85 mmHg or more than 40 mmHg lower than at the initiation of analgosedation for >10 minutes), hypertension (systolic blood pressure >190 mmHg >20 minutes), tachyarrhythmia (ventricular rate >120 for >20 minutes), bradycardia (asystole >10 s or heart rate <40/min for >30 minutes), and/or hypoxaemia (pulse oximetry <85% for >20 minutes).
Comparison of the incidence and prognostic impact of PMI detected by using different troponin assays | 3 days after surgery
  Comparison of the incidence and prognostic impact of PMI detected by using different high-sensitivity cardiac troponin I (hs-cTnI) assays in parallel to the clinical PMI-screening using high-sensitivity cardiac troponin T (hs-cTnT) assays.
Using biomarkers as tools for prediction of major cardiac complications in patients undergoing non-cardiac surgery | 3 days after surgery
  Evaluation of the incremental value of additional cardiovascular biomarkers and continuous vital sign monitoring in the prediction of PMI and other cardiac complications, as well as the prediction of death, and the understanding of the pathophysiology of PMI.

SECONDARY OUTCOMES:
Number of patients with PMI with ischemic symptoms and signs detected in a screening program in high-risk patients undergoing major non-cardiac surgery | 3 days after surgery
  Patients with PMI are evaluated for: presence of chest pain, atypical symptoms, palpitations, dyspnea, edema, or nausea; ST-changes, Q-waves, T-wave abnormalities, new bundle branch block.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Müller, MD, Prof, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No